CLINICAL TRIAL: NCT03685825
Title: Impact of Ophthalmic Surgeon Experience on Early Postoperative Central Corneal Thickness After Cataract Surgery
Brief Title: Impact of Ophthalmic Surgeon Experience on Early Postoperative Central Corneal Thickness
Acronym: CHICA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-14Obs-CHRMT
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Cataract
Keywords: Surgeon experience; Endothelial cell loss
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the impact of surgeon experience on early postoperative central corneal thickness (CCT) in eyes that have undergone phacoemulsification-based cataract surgery.

DETAILED DESCRIPTION:
Cataract surgery is the most commonly performed surgical procedure. Although phacoemulsification is considered a safe method of performing cataract surgery, the risk of endothelial cell loss (ECL) remains.

Given that the surgical technique and speed typically improve with surgeon skill and experience, the purpose of this study was to evaluate the impact of surgeon experience on the occurrence of ECL, as reflected by the presence of corneal edema.

ELIGIBILITY:
Inclusion Criteria:

* Presence of senile cataract
* Age above 50 years
* History of visual acuity regression

Exclusion Criteria:

* Presence of white or Brown cataract
* History of previous ophtalmic surgery
* preexisting corneal pathology (cornea guttata, infectious keratitis or active inflammatory or old)
* Patients who developed intraoperative complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred sixty eyes underwent phacoemulsification-based cataract surgery performed by an experienced surgeon or a less surgically experienced ophtalmic assistant, using the divide-and-conquer or tilt-and-tumble technique for cataractous lens extraction.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2014-03-31 (Actual)

PRIMARY OUTCOMES:
Early postoperative corneal edema | hour 2
  Calculated in micrometers, using pachymetric measurements to estimate central corneal thickness